CLINICAL TRIAL: NCT00147329
Title: A Phase 2, Double-Blind, Placebo-Controlled, Randomized Study To Evaluate the Tolerability, Pharmacokinetics, Pharmacodynamics, and Biologic Activity of MM-093 in Patients With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Safety and Efficacy Study of MM-093 in Patients With Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merrimack Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MM-093-02-200
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2007-02-23 (Estimated); Status verified 2007-02

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

INTERVENTIONS:
Drug: MM-093

SUMMARY:
Merrimack is conducting a research study to see if an experimental drug, called MM-093, is safe and effective in the treatment of psoriasis. MM-093 is a genetically engineered version of a naturally occurring protein called alpha fetoprotein (AFP). Adults normally have very small amounts of AFP in their bloodstream. However, during pregnancy, AFP levels in both the mother and the fetus are much higher than normal. It has been observed that some women with psoriasis and other autoimmune diseases such as rheumatoid arthritis have fewer symptoms during pregnancy, particularly during the third trimester. At this time, the levels of AFP in the blood of the mother and fetus are the highest. This observation led Merrimack to begin examining MM-093 as a potential treatment for psoriasis. This study is designed to further test the safety and effectiveness of MM-093 in patients with psoriasis.

DETAILED DESCRIPTION:
TBA

ELIGIBILITY:
* Aged 18 years and above.
* Understand, sign, and date the written voluntary informed consent form at the screening visit prior to any protocol-specific procedures being performed.
* Have had active plaque psoriasis for at least 6 months.
* Had disease onset at <40 years of age.
* Have had stable disease, as judged by the investigator, for at least 2 months prior to screening.
* Have moderate-to-severe psoriasis that is unresponsive to, or inappropriate for treatment with, topical therapy only.
* Have moderate-to-severe chronic plaque psoriasis as defined by each of the following:
* Have at least 10% of their body covered by disease, AND
* Have a PGA score ≥3, AND
* Have 3 or more lesions that are greater than 2 cm and are easily measured and acceptable for biopsy and photographs.

AND

* Be a candidate for systemic or photo therapy
* Be able and willing to comply with study visits and procedures per protocol.
* Women of childbearing potential must use a medically acceptable means of birth control in an effective manner and agree to continue its use during the study and for 4 weeks after the last dose of study drug. Women who have had a complete surgical hysterectomy or are postmenopausal (absence of menstrual period for at least 1 year) are exempt from this requirement.

Medically acceptable forms of birth control include oral contraceptives, injectable or implantable methods, intrauterine devices, tubal ligation (if performed more than 1 year before screening), or properly used barrier contraception. Additionally, the use of condoms is suggested as an adjunct to the methods previously addressed to protect against sexually transmitted diseases and to provide additional protection against accidental pregnancy.

* Sexually active men must agree to use a medically acceptable form of contraception during the study and continue for 4 weeks after the last dose of study drug.
* Able to store patient kit/cooler containing study drug in a refrigerator at home.
* Use of Investigational biologic agent with in the last 2 months
* Use of Infliximab (Remicade), efalizumab (Raptiva) or alefacept with the last 2 months.
* Use of Investigational drug (NSAID or other small molecule)with in the last 4 weeks
* Use of Cyclosporine, methotrexate, 6-thioguanine or tacrolimus with in the last 4 weeks
* Use of Oral, intramuscular, intravenous or intra-lesional with in the last 4 weeks corticosteroids
* Use of Etanercept (Enbrel) with in the last 4 weeks
* Use of Phototherapy (i.e. UVB, PUVA, excessive sun exposure (or use of tanning booths)with in the last 4 weeks
* Topical therapies for the treatment of psoriasis (The 2 weeks following are allowed: medicated, non-steroidal shampoos; bland emollients, without beta or alpha hydroxyl acids and low potency (Class VI or VII) topical steroids which can only be used on the palms, soles, face and groin.
* Significant concurrent medical diseases including:

Cancer, or a history of cancer, or lymphoproliferative disorder (other than successfully resected cutaneous basal or squamous cell carcinoma) within 5 years before the screening visit.

* Any condition for which participation in this study is judged by the physician to be detrimental to the patient, such as history of significant or unstable cardiac, pulmonary, gastrointestinal, neurological, or psychiatric disease.
* Significant ongoing infection requiring systemic antibiotic, antifungal, antiviral, or any anti-mycobacterial therapy.
* Autoimmune or connective tissue disorder other than chronic active plaque psoriasis, with or without psoriatic arthritis (e.g. Rheumatoid Arthritis, Systemic Lupus Erythematosus, or Scleroderma).
* Other active skin diseases or skin infections (bacterial, fungal, or viral) that may interfere with the evaluation of psoriasis.
* Other forms of psoriatic skin disease including erythrodermic psoriasis, generalized or localized pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new onset guttate psoriasis.
* Grade 2 or above liver function abnormality (i.e. total bilirubin > 1.5 x the upper limit of normal; or aspartate aminotransferase [AST/ SGOT] or alanine aminotransferase [ALT/SGPT] > 2.5 x upper limit of normal).
* Renal disease (including serum creatinine level > 1.5 x the upper limit of normal).
* Any previous history of immunodeficiency syndromes or infection with human immunodeficiency virus (HIV), or a history of hepatitis C or chronic hepatitis B.
* Live viral or bacterial vaccinations within 3 months prior to screening, or planning to receive such vaccinations during the trial, or up to 3 months after the last injection of MM-093.
* Pregnant or breastfeeding women or planning to become pregnant during the study or within 4 weeks after the last dose of study drug.
* Scheduled elective surgery during study participation.
* Participated in any previous clinical trial using MM-093 or have any prior exposure to MM-093.
* History of severe hypersensitivity to goat, sheep or cow milk or products derived from goat, sheep or cow milk (patients who are lactose intolerant are not excluded).
* Any other acute or clinically important condition that the investigator feels would jeopardize the integrity of the study (e.g. a CTCAE grade 2 or above clinical finding or laboratory result).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-09; Study Completion 2006-07

PRIMARY OUTCOMES:
To evaluate safety and tolerability of MM-093 in psoriasis patients.
To evaluate efficacy of MM-093 as measured by percent of patients achieving PASI 50.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Mentor, MD, Principal Investigator; Gerald Krueger, Principal Investigator
Locations (2):
- United States (2):
  - Texas Dermatology Research Institute, Dallas, Texas
  - U. of Utah School of Medicine- Department of Dermatology, Salt Lake City, Utah